CLINICAL TRIAL: NCT00785668
Title: A Phase 1 Safety and Pharmacokinetics Study of AER 001 Administered as a Dry Powder in Asthmatic Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aerovance, Inc. (Industry)
Responsible Party: Aerovance Inc.
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: QGUY/2007/AER 001/-04
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-11

CONDITIONS: Asthma
Keywords: Asthma; Allergy; Interleukin-4; Interleukin-13; IL-4; IL-13; Pharmacokinetics; Safety; Tolerability; Aerovance; dry powder
MeSH Terms: conditions — Asthma; Hypersensitivity; Rhinitis, Allergic | interventions — pitrakinra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AER 001 — 10 mg dry powder administered using a handheld device
  Other Names: AEROVANT, BAY 16-9996, Pitrakinra

SUMMARY:
This is a single centre, single dose pharmacokinetic/safety study in male and female asthmatic subjects. Subjects will receive a single dose of 10 mg of AER 001 administered as a dry powder using a handheld device. The goals of this study are to understand the pharmacokinetics and safety of AER 001 administered as a dry powder in mild to moderate asthmatics.

DETAILED DESCRIPTION:
Study Design

* Single centre, single dose PK/safety study in male and female asthmatic subjects.
* Approximately 10 subjects will be dosed.
* Treatments will be administered by dry powder inhalation using a handheld device
* Subjects will attend the Unit for screening and if eligible return to the Unit on the day of dosing (Day 1). Subjects will be required to stay overnight in the Unit and will be discharged on Day 2.
* On study Day 1, subjects are to receive a single administration of AER 001. N.B. Screening will take place within 28 days prior to administration of AER 001.

Primary objective: To investigate the pharmacokinetics of AER 001 administered as a dry powder in mild to moderate asthmatics.

Secondary objective: To investigate the safety of AER 001 administered as a dry powder in mild to moderate asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females > 18 years.
* Subjects who if female, are not currently pregnant or breast feeding and are using medically acceptable methods of contraception and if male, are themselves and their female partners using medically acceptable methods of contraception.
* Subjects who have a pre study medical history, physical examination, 12 Lead ECG acceptable to the investigator.
* Subjects who have clinical laboratory tests within the reference ranges or clinically acceptable to the investigator.
* Subjects who are negative for HbsAg, hepatitis C antibody and HIV II and I test at screening.
* Subjects who are negative for drugs of abuse at screening and admission.
* Subjects who are negative for alcohol on admission.
* Subjects who have an improvement in FEV1 of >10% following 400 ug salbutamol administration using a spacer device.
* Subjects who have a FEV1 > 70% of predicted at screening and pre dose.
* Subjects who have not received steroid treatment in the prior week.
* Subjects who are non-smokers for at least 3 months prior to screening.
* Subjects who have a < 10 pack year smoking history.
* Subjects who satisfy the Global Initiative in Asthma (GINA, 2002) definition of asthma or have been on treatment for asthma.
* Subjects who have a FEV 1 /FVC ratio >0.65 at screening and pre-dose.
* Subjects with stable, adequately treated medical conditions may be enrolled provided the Principal Investigator does not consider their study participation to place them at increased risk of adverse events. Subjects should continue their concomitant treatments without change during the study.
* Subjects who are able and willing to give written informed consent.

Exclusion Criteria:

* Subjects who do not conform to the above inclusion criteria.
* Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders which would preclude participation.
* Subjects who have a history of relevant drug hypersensitivity.
* Subjects who have a history of alcoholism.
* Subjects who have a history of drug abuse.
* Subjects who consume more than 28 units (male)/ 21 units (female) of alcohol a week.

(unit = 1 glass of wine = 1 measure of spirits = ½ pint of beer)

* Subjects who have acute gastrointestinal symptoms at the time of screening and/or admission (e.g. nausea, vomiting, diarrhoea, heartburn)
* Subjects who have an acute respiratory infection such as influenza at the time of screening and/or admission.
* Female subjects who are pregnant, breast feeding, or not using an acceptable method of contraception. Male subjects whoare not using an acceptable method of contraception or have a partner of child-bearing potential who is not using an acceptable method of contraception.
* Subjects who have used any investigational drug and /or participated in any clinical trial within 3 months of their first dosing.
* Subjects using medication, which in the opinion of the Investigator will affect the outcome of the study.
* Subjects who have donated and/or received any blood or blood products within the previous 3 months prior to first dosing (to review on a case by case basis).
* Subjects who cannot communicate reliably with the investigator.
* Subjects who are unlikely to co-operate with the requirements of the study.
* Subjects who have previously taken AER 001.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-11; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration-time curves will be the primary PK parameter. Maximum observed plasma drug concentrations, time of occurrence of Cmax, the apparent terminal rate constant and corresponding half-life will also be derived. | 24 hours

SECONDARY OUTCOMES:
Safety evaluation will include lung function measurements, blood pressure, heart rate, ECG parameters, clinical laboratory tests (haematology, serum biochemistry, urinalysis, urine and urine microscopy, if required) and adverse events. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MBBS, DCPSA, Principal Investigator — Guy's Drug Research Unit a division of Quintiles Ltd.
Locations (1):
- Guy's Drug Research Unit a division of Quintiles Ltd., London, England, United Kingdom

REFERENCES:
- [Result] Burmeister Getz E, Fisher DM, Fuller R. Human pharmacokinetics/pharmacodynamics of an interleukin-4 and interleukin-13 dual antagonist in asthma. J Clin Pharmacol. 2009 Sep;49(9):1025-36. doi: 10.1177/0091270009341183. PMID 19717725